CLINICAL TRIAL: NCT05252390
Title: Phase 1/2 Safety and Efficacy Study of NUV-868 as Monotherapy and in Combination With Olaparib or Enzalutamide in Adult Patients With Advanced Solid Tumors
Brief Title: NUV-868 as Monotherapy and in Combination With Olaparib or Enzalutamide in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has achieved its objectives.
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NUV-868-01
Record Dates: First submitted 2022-01-28; First posted 2022-02-23 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumor; Ovarian Cancer; Ovary Cancer; Cancer of Ovary; Cancer of the Ovary; Ovary Neoplasm; Pancreatic Cancer; Pancreas Cancer; Cancer of Pancreas; Cancer of the Pancreas; Pancreas Neoplasm; Prostate Cancer; Prostatic Cancer; Cancer of Prostate; Cancer of the Prostate; Prostate Neoplasm; Castrate Resistant Prostate Cancer; Castration Resistant Prostatic Cancer; Castration Resistant Prostatic Neoplasms; Triple-negative Breast Cancer; Triple Negative Breast Cancer; Triple Negative Breast Neoplasms; Breast Cancer; Breast Carcinoma; Cancer of Breast; Cancer of the Breast; Breast Tumor
Keywords: Phase 1; Phase 2; NUV-868; olaparib; enzalutamide; Xtandi; ovarian cancer; pancreatic cancer; metastatic castration-resistant prostate cancer; triple-negative breast cancer; Lynparza; PARP inhibitor; BET inhibitor; BRCA mutation; BRCA1; BRCA2; HRD; HRR deficiency; homologous recombination deficiency
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — olaparib; enzalutamide

STUDY DESIGN:
Intervention Model Description: Sequential assignment will be applied in Phase 1 and Phase 1 b dose escalation cohorts. Parallel assignment will be applied in Phase 1b backfill cohorts and Phase 2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1 Monotherapy (Experimental): NUV-868 will be administered at escalating dose levels until the maximum tolerated dose (MTD) is reached or a recommended Phase 2 dose (RP2D) is determined.
  Interventions: Drug: NUV-868
- Phase 1b Combination: NUV-868 + Olaparib (Experimental): NUV-868 will be administered at escalating dose levels in combination with olaparib until the recommended Phase 2 combination dose (RP2cD) is determined.
  300 mg olaparib will be administered orally twice daily throughout the 28-day cycles of NUV-868.
  Interventions: Drug: NUV-868; Drug: Olaparib
- Phase 1b Combination: NUV-868 + Enzalutamide (Experimental): NUV-868 will be administered daily at escalating dose levels in combination with enzalutamide until the RP2cD is determined.
  160 mg enzalutamide will be administered orally daily throughout the 28-day cycles of NUV-868.
  Interventions: Drug: NUV-868; Drug: Enzalutamide
- Phase 2 Combination: NUV-868 + Olaparib (Experimental): NUV-868 will be administered at the RP2cD.
  Olaparib will be administered at the RP2cD.
  Interventions: Drug: NUV-868; Drug: Olaparib
- Phase 2 Combination: NUV-868 + Enzalutamide (Experimental): NUV-868 will be administered at the RP2cD.
  Enzalutamide will be administered at the RP2cD.
  Interventions: Drug: NUV-868; Drug: Enzalutamide
- Phase 2: NUV-868 Monotherapy (Experimental): NUV-868 will be administered at the RP2D in one arm of a randomized Phase 2 combination (NUV-868 + enzalutamide) cohort.
  Interventions: Drug: NUV-868
- Phase 2: Enzalutamide Monotherapy (Active Comparator): 160 mg enzalutamide will be administered orally daily in one arm of a randomized Phase 2 combination (NUV-868 + enzalutamide) cohort.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: NUV-868 — NUV-868 is an investigational drug for oral dosing.
  Arms: Phase 1 Monotherapy; Phase 1b Combination: NUV-868 + Enzalutamide; Phase 1b Combination: NUV-868 + Olaparib; Phase 2 Combination: NUV-868 + Enzalutamide; Phase 2 Combination: NUV-868 + Olaparib; Phase 2: NUV-868 Monotherapy
Drug: Olaparib — Olaparib
  Other Names: Lynparza
  Arms: Phase 1b Combination: NUV-868 + Olaparib; Phase 2 Combination: NUV-868 + Olaparib
Drug: Enzalutamide — Enzalutamide
  Other Names: Xtandi
  Arms: Phase 1b Combination: NUV-868 + Enzalutamide; Phase 2 Combination: NUV-868 + Enzalutamide; Phase 2: Enzalutamide Monotherapy

SUMMARY:
NUV-868-01 is a first-in human, open- label, Phase 1/2 dose escalation and expansion study in patients with advanced solid tumors. The Phase 1 and 1b portions include patients with advanced solid tumors and are designed to determine the safety and the dose(s) of NUV-868 to be used as monotherapy and in combination with olaparib or enzalutamide for the Phase 2 portion. In Phase 2, NUV-868 in combination with olaparib or enzalutamide will be given to determine the safety and efficacy of these study treatments. One cohort of patients (with enzalutamide-naïve metastatic castration-resistant prostate cancer) will be randomized to receive either NUV-868 monotherapy, enzalutamide monotherapy, or the combination of NUV-868 + enzalutamide. Patients will self-administer NUV-868 orally daily in 28-day cycles as monotherapy in Phases 1 and 2. In Phases 1b and 2, patients will self-administer NUV-868 orally daily in 28-day cycles in combination with olaparib or enzalutamide daily at standard prescribed doses (Phase 1b) or at the recommended Phase 2 combination dose (RP2cD) that is determined in Phase 1b. Patients will be treated until disease progression, toxicity, withdrawal of consent, or termination of the study.

DETAILED DESCRIPTION:
This study was initially planned as a Phase 1/2 study; however, the study stopped early prior to the start of Phase 2.

ELIGIBILITY:
Key Inclusion Criteria For All Phases and Cohorts:

1. Recovered from toxicity to prior anticancer therapy
2. Adequate bone marrow and organ function
3. No known active or symptomatic central nervous system (CNS) disease

Cohort-Specific Inclusion Criteria: In addition to the inclusion criteria listed above, the following criteria apply for enrollment into specific cohorts.

Phase 1 (NUV-868 Monotherapy)

1. Patients with advanced solid tumors that have progressed during or after treatment with approved therapies or for which there is no standard effective therapy available
2. Life expectancy of > 3 months
3. Eastern Cooperative Oncology Group Performance Status ≤ 2
4. Measurable or non-measurable disease

Phase 1b (NUV-868 in Combination With Enzalutamide or Olaparib)

1. Life expectancy of > 3 months
2. Eastern Cooperative Oncology Group Performance Status ≤ 2
3. (Select cohorts only) Measurable disease
4. Patient must be able to read and write sufficiently to document food intake and study drug dosing on the Dosing Diary or must have a caregiver who is willing and able to complete the Dosing Diary with the patient.
5. One of the following tumor types:

   1. Ovarian: Platinum-resistant OR platinum-refractory high grade serous ovarian, fallopian, or primary peritoneal cancer in the relapsed setting
   2. Pancreatic: Pancreatic ductal adenocarcinoma (PDAC) with progression on or after treatment with at least one line of systemic chemotherapy in the advanced setting
   3. Prostate: Histologically confirmed, metastatic adenocarcinoma of the prostate (adenocarcinoma/high grade carcinoma with neuroendocrine features is allowed) with progression on or after treatment with at least one NHT in the metastatic setting
   4. Breast: Triple-negative breast cancer (TNBC) with progression on or after treatment with at least one line of systemic chemotherapy in the advanced setting
   5. Other advanced tumors (only Phase 1b dose escalation, NUV-868 + olaparib): the study Medical Monitor must approve enrollment.
   6. For all tumor types: Patients will be allowed in the study regardless of their BRCA/HRR status.

Phase 2

1. Life expectancy of > 6 months
2. (Select cohorts only): At least one measurable lesion defined by standard criteria
3. Eastern Cooperative Oncology Group Performance Status ≤ 1
4. One of the following tumor types:

   1. Ovarian: Platinum-resistant or platinum- refractory high grade serous ovarian, fallopian, or primary peritoneal cancer in the relapsed setting
   2. Pancreatic: Progression on or after treatment with at least one line of systemic chemotherapy in the advanced setting
   3. Prostate: Histologically confirmed, metastatic adenocarcinoma of the prostate (adenocarcinoma/high grade carcinoma with neuroendocrine features is allowed) with progression on or after treatment with at least one NHT in the metastatic setting
   4. Breast: TNBC with progression on or after treatment with at least one line of systemic chemotherapy in the advanced setting

Key Exclusion Criteria For All Phases and Cohorts:

1. Have received chemotherapy, hormonal therapy (except for ongoing luteinizing hormone-releasing hormone [LHRH] analogs in male patients and premenopausal women), radiation, or biological anticancer therapy within 14 days prior to the first dose of NUV-868.
2. Received treatment with an investigational agent for any indication within 14 days for non-myelosuppressive agent, or within 21 days or < 5 half-lives (whichever is longer) for myelosuppressive agent, prior to the first dose of study treatment.
3. Requires medications that are known to be strong (or moderate for olaparib) inducers and/or strong (or moderate for olaparib) inhibitors of CYP3A4/5 enzymes.
4. Female patients who are pregnant of breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Phase 1 Monotherapy Dose Escalation: Safety and tolerability of NUV-868 to determine the recommended Phase 2 dose (RP2D) | During the DLT period (28 days)
  Incidence of dose-limiting toxicities (DLTs)
Phase 1b Dose Escalation, NUV-868 + Olaparib: Safety and tolerability of NUV-868 in combination with olaparib to determine the recommended Phase 2 combination dose (RP2cD) | During the DLT period (28 days)
  Incidence of DLTs
Phase 1b Dose Escalation, NUV-868 + Olaparib: Pharmacokinetic (PK) profiles of NUV-868 and olaparib when administered in combination | Days 1, 8, and 29
  NUV-868 and olaparib combination PK
Phase 1b Dose Escalation, NUV-868 + Enzalutamide: Safety and tolerability of NUV-868 in combination with enzalutamide to determine the RP2cD | During the DLT period (28 days)
  Incidence of DLTs
Phase 1b Dose Escalation, NUV-868 + Enzalutamide: Pharmacokinetic (PK) profiles of NUV-868 and enzalutamide when administered in combination | Days 1, 8, and 57
  NUV-868 and enzalutamide combination PK
Phase 2, NUV-868 + Olaparib: Change from Baseline in Tumor Imaging | Every 8 weeks during the first 24 weeks and then every 12 weeks, up to an average of 12 months (end of treatment)
  ORR per standard criteria
Phase 2, NUV-868 + Olaparib: Change from Baseline in PSA measurements | Every 4 weeks throughout study treatment, up to an average of 12 months (end of treatment)
  PSA50 response rate per standard criteria; only for patients with prostate cancer
Phase 2, NUV-868 + Enzalutamide in Enzalutamide-Naïve Metastatic Castrate-Resistant Prostate Cancer (mCRPC): Time from First Dose to Disease Progression | Every 8 weeks during the first 24 weeks and then every 12 weeks, up to an average of 12 months (end of treatment)
  Radiographic progression-free survival (rPFS) per standard criteria
Phase 2, NUV-868 + Enzalutamide in Enzalutamide-Resistant mCRPC: Response to Study Treatment | Every 4-12 weeks (time points vary depending on the type of response being evaluated) throughout study treatment, up to an average of 12 months (end of treatment)
  Composite response rate (CRR: radiologic response, PSA50 response, and/or circulating tumor cell response) per standard criteria
Phase 1b Food Effect Substudy: Effect of Food on the Pharmacokinetics (PK) of NUV-868 | Pre dose and 24 hours after the first and second doses of NUV-868, 7 days apart
  NUV-868 PK parameters in fed and fasted states

CONTACTS AND LOCATIONS:
Locations (22):
- United States (17):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Ellison Institute of Technology, Los Angeles, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Laura & Isaac Perlmutter Cancer Center - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (5):
  - Macquarie University Hospital, North Ryde, New South Wales
  - Calvary Mater Hospital Newcastle, Waratah, New South Wales
  - Cabrini Hospital Malvern, Malvern, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia